CLINICAL TRIAL: NCT04611386
Title: Bursa Postgraduate Hospital
Brief Title: The Effect of Contrast Agents on the Anticoagulant Properties of Oral Factor Xa Inhibitors
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: Bursa Yüksek İhtisas EAH
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Contrast Agents and Oral Factor Xa Inhibitor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- rivaroxaban group: 20 rivaroxaban using patients
  Interventions: Drug: computerized tomography
- apixaban group: 20 apixaban using patients
  Interventions: Drug: computerized tomography
- edoxaban group: 20 edoxaban using patients
  Interventions: Drug: computerized tomography
- control group: 5 control group patients
  Interventions: Drug: computerized tomography

INTERVENTIONS:
Drug: computerized tomography — Anti Factor Xa level

SUMMARY:
The aim of this study is to evaluate the effect of iohexol as a contrast agent on the anticoagulant activity of oral factor Xa inhibitors.

DETAILED DESCRIPTION:
The study included 65 people who underwent contrast computerized tomography (CT). The study patients were divided into 4 groups. Patients in group 1 were using rivaroxaban (20 patients), patients in group 2 were using apixaban (20 patients), patients in group 3 were using edoxaban (20 patients), and group 4 was the control group (5 volunteers). Iohexol (60 ml) was used as a contrast agent. Two tubes were used to collect 2 ml of blood from the patients at 4 hours after the drug dose (rivaroxaban, apixaban, or edoxaban) and 1 hour after the contrast CT (CT was performed 3 hours after the drug was taken). In the control group, at any time and 1 hour after contrast CT, 2 tubes of 2 ml of blood were collected. The anticoagulant properties of rivaroxaban, apixaban, and edoxaban were evaluated using anti-factor Xa levels.

ELIGIBILITY:
Inclusion Criteria:

1. the use of oral factor Xa inhibitors (patients with nonvalvular AF and CHA2DS2-VASc Score ≥2),
2. age of 21-80 years,
3. no contraindications for anticoagulation use,
4. GFR greater than 30,
5. volunteering to participate in the study, and
6. patients who needed to use contrast agent (iohexol) for CT examination. -

Exclusion Criteria:

1. coagulopathy,
2. severe hepatic insufficiency,
3. chronic systemic or inflammatory diseases,
4. patients lighter than 60 kg,
5. malignancy,
6. creatinine value above 1.5 mg/dl, and
7. not providing consent to participate in the study -

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study prospectively included 65 people who underwent contrast computerized tomography (CT). The CT indications were thoracic aortic dilatation, chronic obstructive pulmonary disease, abdominal aortic dilatation, chronic abdominal pain.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Anti Factor Xa level | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavlan B, Ari S, Ari H, Camci S, Melek M, Bozat T. The effect of contrast agents on the anticoagulant properties of oral factor Xa inhibitors. Acta Radiol. 2023 Feb;64(2):588-595. doi: 10.1177/02841851221081474. Epub 2022 Mar 16. PMID 35296141